CLINICAL TRIAL: NCT02333591
Title: Effect of Intact GLP-1 (7-36) and GLP-1 Metabolite (9-36) on Coronary and Peripheral Vascular Function in Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mette Zander (Other)
Collaborators: Hvidovre University Hospital (Other)
Responsible Party: Sponsor-Investigator, Mette Zander, MD, PhD, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: MZ02; 2013-001240-64 (EudraCT Number)
Record Dates: First submitted 2015-01-06; First posted 2015-01-07 (Estimated); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Coronary Microvascular Dysfunction
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- GlucagonLikePeptide-1 (7-36) (Active Comparator): GLP-1 (7-36) is diluted in saline and human serum albumin. Plasma levels of GLP-1 (7-36) are rapidly raised and then maintained stable with 5,91 pmol/kg/min (0-2 min) reduced to 2,53 pmol/kg/min (2-4 min) reduced to 2,34 pmol/kg/min (4-6 min) reduced to 2,2 pmol/kg/min (6-8 min) reduced to 2,02 pmol/kg/min (8-10 min) and then maintained stable for 2½ hours with 1.5 pmol/kg/min.
  A DPP-IV inhibitor - Januvia 100 mg is given the evening before and ½ an hour before the infusion is started.
  Interventions: Drug: Saline
- GlucagonLikePeptide-1 (9-36) (Active Comparator): GLP-1 (9-36) is diluted in saline and human serum albumin. Plasma levels of GLP-1 (9-36) are rapidly raised and then maintained stable with 5,91 pmol/kg/min (0-2 min) reduced to 2,53 pmol/kg/min (2-4 min) reduced to 2,34 pmol/kg/min (4-6 min) reduced to 2,2 pmol/kg/min (6-8 min) reduced to 2,02 pmol/kg/min (8-10 min) and then maintained stable for 2½ hours with 1.5 pmol/kg/min
  Interventions: Drug: Saline
- NaCl (Placebo Comparator): Saline is infused with a flow rate of 240 ml/h for 10 min and then reduced to 86 ml/h for 2½ hours.
  Interventions: Drug: GlucagonLikePeptide-1 (7-36); Drug: GlucagonLikePeptide-1 (9-36)

INTERVENTIONS:
Drug: GlucagonLikePeptide-1 (7-36) — Diluted in saline and human serum albumin, then infused intravenously for 2,5 hours.
  Arms: NaCl
Drug: GlucagonLikePeptide-1 (9-36) — Diluted in saline and human serum albumin, then infused intravenously for 2,5 hours.
  Arms: NaCl
Drug: Saline — Infused intravenously for 2,5 hours.
  Other Names: NaCl, Placebo
  Arms: GlucagonLikePeptide-1 (7-36); GlucagonLikePeptide-1 (9-36)

SUMMARY:
GLP-1 is an agent for treatment of type 2 diabetes and may have protective effects on the cardiovascular system. The mechanism is complex and there seems to be a dual function with intact GLP-1 (7-36), acting through the GLP-1 receptor, and the GLP-1 (9-36) metabolite acting independently of the GLP-1 receptor.

Coronary flow reserve (CFR) is the ratio of flow through the coronary arteries during stress to during rest and it reflects coronary microcirculation. Impaired CFR is a strong predictor of poor prognosis of cardiovascular disease.

The aim of the study is to investigate the acute effects of GLP-1 on coronary microcirculation and endothelial function in adults with obesity.

DETAILED DESCRIPTION:
Several studies have shown beneficial effects of glucagon-like-peptide-1 (GLP-1) on the cardiovascular system. Native GLP-1 is secreted from L-cells in the intestine as GLP-1(7-36) 1 but is rapidly metabolised by the ubiquitous enzyme dipeptidyl-peptidase-4 (DPP4) to the metabolite GLP-1(9-36). However, the physiological effect of GLP-1 on the cardiovascular system is complex and there seems to be a dual function with intact GLP-1 (7-36), acting through the GLP-1 receptor, and the GLP-1 (9-36) metabolite acting independently of the GLP-1 receptor.

The aim of the study is to investigate the acute effects of intact GLP-1 and GLP-1 metabolite on coronary microcirculation and endothelial function in adults.

Method 20 adults with obesity are recruited to a double-blind randomized cross-over study.

The first 10 included adults will receive 2½ hours infusion of intact GLP-1 (7-36) together with a DPP-IV inhibitor and 2½ hours infusion of saline, on two separate occasions. The infusions will be given in randomized order with a minimum of 24 hours washout period.

The next 10 included adults will receive 2½ hours infusion of GLP-1 (9-36) metabolite and 2½ hours infusion of saline. These will also be given in randomized order with a minimum of 24 hours washout period. Endothelial function and CFR will be measured before and after one, respectively two, hours of infusion.

The effect of GLP-1 infusions on microvascular function is evaluated by coronary flow reserve (CFR), the ratio between echocardiographic measured coronary flow velocity in LAD during adenosine induced myocardial hyperaemia and rest. The effect on endothelial function is assessed by flow mediated dilation (FMD).

ELIGIBILITY:
Inclusion Criteria:

* Age 35-70 years
* BMI > 25 kg/m2.
* Central obesity (measured by waist circumference, defined as ≥ 94cm for men and ≥ 80 cm for women)
* Non smokers (6 months abstinent is required)
* Normal creatinine
* For fertile women; negative pregnancy test and use of safe anticonception.
* Speak and understand Danish or English
* Mental ability to follow and understand the study

Exclusion Criteria:

* Known Diabetes
* Known hypertension (untreated hypertension ≤ 160/100 at inclusion is accepted)
* Haemoglobin < 6.5 mmol/l
* Allergy towards Januvia or Exenatide, Adenosin or Glycerylnitrate
* Documented significant stenosis of the left anterior descending artery (LAD) at coronary angiography or CT-angiography or regional dysfunction documented during dipyridamol stress-echocardiography. If stress test at baseline shows significant stenosis the patient will be excluded from the study.
* Pregnancy
* Severe asthma
* Active cancer, severe co-morbidity with limited life-expectancy, severe hepatic co-morbidity, chronic alcohol abuse, atrial fibrillation, chronic or previous acute pancreatitis, inflammatory bowel disease.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-07; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Coronary Flow Reserve | At baseline and after 2 hours of infusion
  Coronary flow reserve (CFR) reflects microvessel coronary function and is the ratio between echocardiographic measured coronary flow velocity in LAD during adenosine induced myocardial hyperaemia and rest.
  The outcome is measured at every infusion/intervention (4 times).

SECONDARY OUTCOMES:
Endothelial function (Assessed by Flow Mediated Dilation) | At baseline and after 1 hour of infusion
  Assessed by Flow Mediated Dilation (FMD) The outcome is measured at every infusion/intervention (4 times).

CONTACTS AND LOCATIONS:
Overall Officials: Mette Zander, PhD, MD, Principal Investigator — Department of Endocrinology, Bispebjerg University Hospital
Locations (1):
- Department of Research in Endocrinology, Bispebjerg University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided